CLINICAL TRIAL: NCT03398564
Title: Efficacy of Ultrasound-Guided Erector Spinae Plan Block on Postoperative Pain After Laparoscopic Cholecystectomy Under General Anesthesia. Randomized, Controlled Trial
Brief Title: Erector Spinae Plan Block for Postoperative Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al Jedaani Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1/12
Record Dates: First submitted 2017-12-29; First posted 2018-01-12 (Actual); Last update posted 2018-12-26 (Actual); Status verified 2018-10

CONDITIONS: Postoperative Pain
Keywords: Erecror Spinae Plan Block; postoperative pain; Laparoscopic cholecystectomy
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Control) (Placebo Comparator): ultrasound guided Bilateral Erector Spinae Plan Block using isotonic saline
  Interventions: Procedure: Erector Spinae Plan Block
- Group II (ESP) (Active Comparator): ultrasound guided Bilateral Erector Spinae Plan Block with bupivacaine 0.25%
  Interventions: Procedure: Erector Spinae Plan Block
- Group III(OSTAP) (Active Comparator): Ultrasound-guided bilateral oblique subcostal TAP block
  Interventions: Procedure: Oblique subcostal TAP

INTERVENTIONS:
Procedure: Erector Spinae Plan Block — The trocar site incision was done 15 minutes after the block in the three groups. The skin was disinfected with chlorhexidine solution, and the high-frequency transducer was isolated with a sterile disposable plastic cover and gel. The patient was placed in lateral position. A high-frequency linear ultrasound probe was placed longitudinally lateral to the T8 spinous process by 3 cm. After identification of the 3 muscles superficial to the hyperechoic transverse process shadow as follows: trapezius, rhomboid major, and erector spinae. The needle was introduced in a cephalo-caudal orientation. The needle tip was positioned fascial plane between rhomboid major and erector spinae muscles. Hydrodissection by 1-2 ml of normal saline to visualize the plan, then deposition of local anesthetic was done. A total of 20 mL of 0.25% bupivacaine was injected here. The same procedure was repeated on the other side.
  Arms: Group I (Control); Group II (ESP)
Procedure: Oblique subcostal TAP — ultrasound-guided bilateral oblique subcostal TAP block with bupivacaine 0.25% (20ml on each side)
  Arms: Group III(OSTAP)

SUMMARY:
Laparoscopic cholecystectomy is a widely employed procedure in ambulatory surgery. Pain after laparoscopic cholecystectomy arises significantly from port site incisions in the anterior abdominal wall. Innervation of the anterior abdominal wall is segmentally supplied by pain afferents in the plane of fascia between transversus abdominis and the internal oblique muscles. Opioids analgesia is used to control postoperative pain, but it carries the risk of increased nausea and vomiting, ileus and sedation that may delay hospital discharge.

Several techniques have been tried as.neuroaxial narcotics, intraperitoneal lavage of local anesthetic and transversus abdominis plan (TAP) block and successfully reduced opioid use and improve postoperative analgesia.

The ultrasound-guided erector spinae plan(ESP) block is a recently described technique which produces reliable unilateral analgesia at thoraco-lumbar dermatomes. ESP block carries the advantages of being simple, safe, easily recognizable by ultrasound, and a catheter can be threaded to extend the duration of analgesia.

Few case series reported the efficacy of (US)-guided ESP blocks in reducing postoperative pain and opioids consumption.

Because of that, the investigators aimed to test the hypothesis that US-guided ESP blocks can decrease opioid consumption during the first 24 h after of laparoscopic cholecystectomy in comparison with the conventional systemic analgesia.

ELIGIBILITY:
Inclusion Criteria:

* 60 ASA I- II adult patients
* 20-60 years old
* elective laparoscopic cholecystectomy
* Body mass index (BMI) less than 35
* Port sites at or above thoracic T 10 dermatome

Exclusion Criteria:

* Allergy to amino-amide local anesthetics
* Presence of coagulopathy
* Local skin infection at the needle puncture sites
* Preoperative chronic dependence upon opioid and NSAID medications
* Liver or renal insufficiency
* History of psychiatric or neurological disease
* Deafness
* previous open surgery that need the conversion of laparoscopic to open surgery or manipulations more than expected with more tissue trauma
* American Society of Anesthesiologists (ASA) above Class II

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2018-01-10 (Actual); Primary Completion 2018-11-30 (Actual); Study Completion 2018-11-30 (Actual)

PRIMARY OUTCOMES:
Morphine consumption | 24 hours postoperatively.
  It was calculated as equivalent morphine dose to the opioid analgesia consumed

SECONDARY OUTCOMES:
Quality of analgesia | Every 2 hours for 24 hours postoperatively
  comparing visual analog scores (VAS) every two hours after surgery
The intraoperative fentanyl | 2 hours
  (µg) required during surgery
equivalent morphine dose in the recovery unit (PACU) | one hour
  equivalent morphine dose in the recovery unit (PACU)
Erector spinae plan block complications | 24 hours postoperative
  local anesthetic systemic toxicity, vascular injury, and intravascular injection of local anesthetic

CONTACTS AND LOCATIONS:
Locations (1):
- Al Jedaani group of hospitals, Jeddah, Meccah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ibrahim M. Erector Spinae Plane Block in Laparoscopic Cholecystectomy, Is There a Difference? A Randomized Controlled Trial. Anesth Essays Res. 2020 Jan-Mar;14(1):119-126. doi: 10.4103/aer.AER_144_19. Epub 2020 Feb 3. PMID 32843804